CLINICAL TRIAL: NCT06536660
Title: Development and Application of Biodegradable Magnesium Bone Plate and Screw Fixation in Jaw Surgery
Brief Title: Biodegradable Magnesium Bone Plate and Screw Fixation in Jaw Surgery
Acronym: MgJawSurgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Leung Yiu Yan, Clinical Professor in Oral and Maxillofacial Surgery, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 24-175
Record Dates: First submitted 2024-06-26; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Orthognathic Surgical Procedures
Keywords: Biodegradable Magnesium Bone Plate; Screw Fixation; Jaw Surgery; Orthognathic Surgical Procedures
MeSH Terms: interventions — Orthognathic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnesium bone plate and screw fixation in jaw surgery (Experimental)
  Interventions: Procedure: Magnesium bone plate and screw fixation in jaw surgery

INTERVENTIONS:
Procedure: Magnesium bone plate and screw fixation in jaw surgery — Participants will undergo jaw surgery based on their clinical indications. High-purity magnesium bone plates and screws will be used for internal fixation during the surgical procedure.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of using high-purity magnesium bone plates and screws for internal fixation in jaw surgery. The investigators aim to assess whether these biodegradable magnesium devices promote normal bone healing and functional recovery while ensuring the safety of patients undergoing dentoalveolar surgery, fracture fixation, orthognathic surgery, or craniofacial reconstruction. The hypotheses are:

1. High-purity magnesium bone plates and screws are effective in bone fixation, promoting normal bone healing and functional recovery in jaw surgery.
2. High-purity magnesium bone plates and screws are safe in jaw surgery in terms of local side effects and systemic safety.

Participants will undergo jaw surgery based on the clinical indications. High-purity magnesium bone plates and screws will be used for internal fixation during the surgical procedure. Participants will be followed up at 1 week, 3 weeks, 6 weeks, 3 months, 6 months, 1 year, and 2 years after surgery to assess wound healing, functional recovery, and any side effects. If any side effects occur or deemed necessary, participants may be followed up for a longer period. During postoperative follow-up visits, X-ray or CBCT/CT imaging will be conducted routinely or when clinically indicated.

DETAILED DESCRIPTION:
Bone plate and screw fixation is a well-recognized system for internal fixation in jaw surgery, encompassing fracture fixation, orthognathic surgery, and craniofacial reconstruction. Along the development, titanium and its alloys have become the predominant materials for internal fixation, owing to their exceptional mechanical properties and biocompatibility. However, titanium has certain drawbacks, such as excessive rigidity compared to bone, which can result in stress shielding and subsequent bone resorption. Additionally, titanium plate and screw fixation is intended for temporary mechanical support during bone healing and may necessitate removal via a secondary surgery following bone healing, thereby increasing healthcare burdens. If left in situ, titanium can interfere with X-ray imaging due to beam-hardening effects.

In an effort to address the limitations of titanium fixation, researchers have been exploring the development of alternative materials for internal fixation. Bioresorbable systems utilize biodegradable materials for bone plate and screw fixation, thus eliminating the need for a secondary surgery for hardware removal. These biodegradable systems avoid long-term issues associated with stress shielding or X-ray scattering. Commercially available biodegradable osteosynthesis materials include high-molecular-weight polymers such as poly(lactic acid) (PLA), polyglycolic acid (PGA), and poly(lactic-co-glycolic acid) copolymer (PLGA). However, these biodegradable polymers exhibit insufficient mechanical strength, necessitating increased dimensions and resulting in a bulky volume that may impede application. Moreover, the suboptimal biocompatibility can provoke foreign body reactions and hinder normal bone healing. Lastly, controlling the biodegradation rates of polymers is challenging, which may surpass normal bone healing and lead to postoperative complications such as malunion or nonunion.

In recent years, magnesium has emerged as a promising biodegradable metal for internal fixation, as demonstrated by numerous research studies. Magnesium exhibits mechanical properties more closely aligned with human bone than the rigid titanium or stainless-steel materials, effectively mitigating the drawbacks of stress shielding and X-ray scattering. In vivo, magnesium plates and screws gradually dissolve, releasing magnesium ions and hydrogen gas. Magnesium ions, essential to the human body, can be metabolized without causing harm. The accumulation of hydrogen gas in tissues may result in temporary swelling or discomfort, which typically resolves as the gas dissipates over time. More importantly, magnesium has demonstrated remarkable bioactivity in promoting bone regeneration, sparking a surge of interest in basic biomechanical research. Its exceptional bioactivity has even been demonstrated in challenging clinical situations. Consequently, the unique and superior properties of magnesium have positioned it as a promising next-generation biomedical implants for internal fixation in humans.

The application of magnesium-based materials in bone surgery can be traced back to 1906, and recent advancements have led to the development of biodegradable internal fixation devices by companies like Synntellix AG (Germany) and U&I Corporation (South Korea) [7]. These fixation systems, including MAGNEZIX® (Mg-Y-Re-Zr alloy screws) and RESOMET™ (Mg-Ca-Zn alloy screws), have shown promising results in various clinical studies across multiple countries, treating conditions such as hallux valgus, osteonecrosis of the femoral head, and distal radius fractures. However, given the potential health risks of alloy elements to patients, Chinese research teams have been committed to the development of high-purity magnesium for internal fixation purposes.

Numerous human clinical studies utilizing high-purity magnesium have been successfully conducted in China. In 2015, Yu et al. employed high-purity magnesium screws for the fixation of vascularized bone grafts in young adults with displaced femoral neck fractures. Over a 16-month follow-up period, patients achieved satisfactory results in the Harris hip score, a functional index, and experienced a lower incidence of complications such as avascular necrosis and nonunion. In 2016, Zhao et al. implemented high-purity magnesium screws in a clinical trial to fix vascularized bone grafts in osteonecrosis of the femoral head. Within a 12-month follow-up period, patients treated with magnesium screws demonstrated higher satisfactory results in functional scores and reduced bone graft displacement. The serum levels of magnesium remained within the normal physiological range, and potential adverse effects induced by magnesium degradation products were absent. In 2019, Chen et al. utilized high-purity magnesium screws to fix vascularized bone grafts for trauma-induced femoral head necrosis in a case report. Satisfactory outcomes were achieved in terms of functional recovery, and the magnesium screws gradually degraded over more than two years without any noticeable side effects.

Despite its potential, magnesium-based fixation faces challenges in orthopedics due to its relatively weak mechanical strength when used in weight-bearing areas, and no clinical trials have been conducted in such cases thus far. Theoretically, fixation in the hip joint area must withstand forces exceeding 2000N, or three times the body weight, which may increase during functional mobilization. Researchers have been exploring coating strategies to decelerate the in vivo degradation of magnesium, thereby extending the mechanical support for adequate orthopedic healing. They are also investigating metallurgical techniques to enhance the mechanical strength of magnesium fixation devices. Conversely, jaw surgeries may benefit from magnesium-based fixation due to their comparatively lower force-loading requirements compared to limb or spine fixation. The normal forces for the mandible are approximately 400N, which decrease to 115N at one week and 250N at six weeks after internal reduction. Consequently, magnesium fixation holds promise for successful application in jaw surgery.

Nonetheless, owing to limited clinical research in this domain, considerable efforts are needed to thoroughly comprehend the benefits of magnesium-based materials in jaw surgery and to establish novel surgical protocols for their implementation. This study seeks to investigate the application of magnesium for bone fixation in jaw surgery and to comprehensively assess the surgical outcomes. The study will contribute to a deeper understanding of using magnesium as internal fixation in jaw surgery and is expected to pave the way for new surgical protocols utilizing biodegradable fixation. Ultimately, this could lead to improved patient outcomes and a reduction in healthcare burdens.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18 years of age or older.
2. Participants must have confirmed indications for jaw surgery with internal fixation, such as alveolar onlay bone grafting, fracture fixation, orthognathic surgery, or reconstructive surgery.
3. Participants should have adequate bone quality and sufficient bone volume to support the placement of magnesium bone plates and screws.
4. Participants must provide written informed consent, indicating their understanding of the potential risks and benefits of magnesium bone plate and screw fixation.

Exclusion Criteria:

1. Participants with certain medical conditions that may affect bone healing or increase the risk of complications, such as uncontrolled diabetes, severe osteoporosis, multiple myelomas, or active bone infections.
2. Participants with medical conditions that may exacerbate or predispose them to systemic side effects of magnesium implants, thus contraindicating their use, should be excluded. These conditions include chronic kidney disease, hypermagnesemia, severe electrolyte imbalances, severe heart disease (especially in those with a history of arrhythmias or heart failure), myasthenia gravis, abnormal thyroid functions, hyperparathyroidism, and adrenocortical insufficiency.
3. Participants with known allergies or hypersensitivity to magnesium.
4. Participants with an ASA score of 3 or above, indicating a higher risk for general anesthesia.
5. Participants who are pregnant or breastfeeding.
6. Participants deemed unlikely to comply with the study protocol, such as attending follow-up appointments or adhering to post-operative care instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2027-08-15 (Estimated); Study Completion 2028-08-15 (Estimated)

PRIMARY OUTCOMES:
The efficacy of using high-purity magnesium bone plate and screw fixation in jaw surgery | 1 week - 2 years
  Efficacy is defined as the rate of successful bone healing and intended functional recovery of the jaw after surgery. Efficacy will be evaluated by clinical assessment and radiological assessment in terms of normal bone healing and functional recovery. Patients will be followed up at 1 week, 3 weeks, 6 weeks, 3 months, 6 months, 1 year, and 2 years after surgery. The occlusal function will be evaluated by the occlusal alignment and the resumption of normal diet. The bone structure will be assessed using plain X-ray immediately after surgery, and at 3 months, 6 months, 1 year, and 2 years post-surgery. CBCT/CT will also be performed to evaluate bone healing and potential complications immediately after surgery (serving as baseline reference), and at 3 months and 1 year after surgery. If CBCT/CT is taken, then plain X-ray will be omitted. The postoperative X-ray schedules represent standard procedures at our center for patients undergoing internal fixation.

SECONDARY OUTCOMES:
Magnesium degradation | 1 week - 2 years
  Magnesium degradation refers to the process of magnesium dissolving or corroding over time in body fluids, eliminating the need for additional surgeries to remove the implant. The degradation rate of magnesium will be monitored over time to ensure a close match with bone healing, providing sufficient support and fixation throughout the healing process. Additionally, the production and retention of hydrogen gas will be monitored during the degradation process, as excessive hydrogen gas accumulation could lead to temporary swelling or discomfort in surrounding tissues, which will be counted as local side effects if clinically symptomatic.
Local side effects | 1 week - 2 years
  Local side effects or complications, such as emphysema, infection, implant rejection, screw loosening, or delayed healing, will be closely monitored.
Systemic side effects | 1 week - 2 years
  Magnesium ions should be metabolized without causing detrimental effects on vital organs or overall health; however, a sudden release of magnesium ions could potentially result in hypermagnesemia, leading to cardiovascular complications or neurological disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Yiu Yan Leung, Principal Investigator — The University of Hong Kong